CLINICAL TRIAL: NCT04493801
Title: Incidence of Rhinological Morbidities During Endonasal Pituitary Surgery, With or Without Nasoseptal Flap
Acronym: HLNS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: HLNS ( 29BRC18.0257)
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-06

CONDITIONS: Surgery--Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with nasoseptal flap: patient who undergo a pituitary gland surgery with nasoseptal flap
- without nasoseptal flap: patient who undergo a pituitary gland surgery without nasoseptal flap

SUMMARY:
Determine and compare prospectively the incidence of rhinological adverse events during pituitary surgery with or without nasoseptal flap

ELIGIBILITY:
Inclusion Criteria:

* to be over 18 years old
* to be operated on for pituitary surgery
* to have express no objection to the study

Exclusion Criteria:

* refusal to participate in the study
* pregnant women
* to be Under the age of 18
* not being able to understand and accept participation in the study
* to have a life expectancy of less than a year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who undergoing a pituary gland surgery
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
post operative epistaxis | during two month after surgery
  no epistaxis - begnin epistaxis - severe epistaxis.
post operative rhinoliquorrhea | during two month after surgery
  physical examination and symptomatic rhinorrhea

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France